CLINICAL TRIAL: NCT07122323
Title: Comparison of Robotic Arm-assisted THA and Conventional Manual THA in Patients With Legg-Calvé-Perthes Disease: a Prospective Cohort Study
Brief Title: Robotic Arm-assisted THA Vs. Conventional THA in Legg-Calvé-Perthes Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiang Zhao, MD, Principal Investigator, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1100
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Legg-Calvé-Perthes Disease
Keywords: MAKO; Legg-Calvé-Perthes disease; flat hip
MeSH Terms: conditions — Legg-Calve-Perthes Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional total hip replacement (Active Comparator): applying conventional total hip replacement in patients with Legg-Calvé-Perthes disease
  Interventions: Procedure: conventional total hip replacement
- robotic arm-assisted total hip replacement (Experimental): applying robotic arm-assisted total hip replacement in patients with Legg-Calvé-Perthes disease
  Interventions: Procedure: robotic arm-assisted total hip replacement

INTERVENTIONS:
Procedure: robotic arm-assisted total hip replacement — using robotic total hip replacement in patients with Legg-Calvé-Perthes disease
  Arms: robotic arm-assisted total hip replacement
Procedure: conventional total hip replacement — applying conventional total hip replacement in patients with Legg-Calvé-Perthes disease
  Arms: conventional total hip replacement

SUMMARY:
Flat hip, also called Legg-Calvé-Perthes disease, is clinically characterized by flattened femoral head, shortened femoral neck, and a center of rotation of the femoral head lower than the apex of the greater trochanter. Joint replacement is difficult, with high intraoperative and postoperative complications. Especially, issues such as unequal limb length, postoperative dislocation, postoperative neurological damage, and prosthesis impact have always plagued clinical practice.

The robotic arm-assisted joint replacement technology has been developed and clinically applied for over 10 years, but it was not until the past 3 years that it began to be widely implemented worldwide. Existing research data indicates that robotic arm-assisted joint replacement technology can significantly improve the placement of prostheses and lower limb force lines in patients, and improve their short-term clinical prognosis. However, its application in complex hips, such as flat hip, is limited. More relevant literature is needed to further enrich people's understanding of this technology. In theory, robot assisted technology can solve many challenges faced in flat hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* patients with Legg-Calvé-Perthes disease and accept total hip replacement in our center

Exclusion Criteria:

* infection, cannot complete follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2027-07-28 (Estimated); Study Completion 2027-07-28 (Estimated)

PRIMARY OUTCOMES:
inclination angle | 2 days after surgery
  The inclination angle in total hip replacement (THR), also called the abduction angle , refers to the angle at which the acetabular cup component is tilted relative to the horizontal plane when viewed on an anteroposterior (AP) pelvic X-ray.
anteversion angle | 2 days after surgery
  The anteversion angle in total hip replacement (THR) refers to the forward tilt (rotation) of the acetabular cup component around its vertical axis. It determines whether the cup's opening faces more forward or backward relative to the pelvis.
Hospital for Special Surgery Score score (HSS score) | before the surgery, 1 week after surgery, 1 month after surgery, 6 months after surgery, 1 year after surgery
  The maximum values is 100, and the minimum value is 0. Higher scores means a better outcome.

SECONDARY OUTCOMES:
operation duration | during the operation
  The operation duration (also called operative time or surgical time ) refers to the total time taken to complete a surgical procedure.
blood loss | during the operation
  The amount of blood loss during the surgery.
Visual Analogue Scale score (VAS score) | before the surgery, 1 week after surgery, 1 month after surgery, 6 months after surgery, 1 year after surgery
  The maximum value is 10, and the minimum value is 0. Lower score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No